CLINICAL TRIAL: NCT03254875
Title: Individually Tailored Rehabilitation After Breast Cancer
Brief Title: Rehabilitation After Breast Cancer
Acronym: REBECCA II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Cancer Society (Other)
Collaborators: Rigshospitalet, Denmark (Other); Copenhagen University Hospital at Herlev (Other)
Responsible Party: Principal Investigator, Christoffer Johansen, Professor, DMSc, Danish Cancer Society
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: REBECCA II
Record Dates: First submitted 2017-07-31; First posted 2017-08-21 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer
Keywords: Breast cancer, Psychosocial intervention
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: During a 2-year period, 758 patients newly diagnosed with breast cancer will be screened for inclusion at the Section of Breast Surgery at Rigshospitalet, Copenhagen. Of these 324 participants enter the RCT and are randomized in a computer-generated sequence of 1:1 to the intervention (nurse-navigation) or control group (standard care). A total of 432 participants will enter an observational questionnaire study. All participants are followed for 1,5 years.
Who Masked: Outcomes Assessor
Masking Description: Intervention status will be blinded in analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Individually tailored nurse navigation
  Interventions: Behavioral: Individually tailored nurse navigation
- Control (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Individually tailored nurse navigation — The intervention consists of systematic report of symptoms to the nurse and up to six individual, manual-based, face-to-face or telephone nurse navigator sessions depending on individual needs.
  Arms: Intervention

SUMMARY:
The aim of the study is to evaluate whether a screening-based individually tailored nurse navigator intervention compared to standard care significantly reduce psychological and physical symptoms among women being treated for breast cancer who had moderate-to-severe distress (score ≥ 7 on the distress thermometer).

DETAILED DESCRIPTION:
During a 2-year period, 758 patients newly diagnosed with breast cancer will be screened for inclusion at the Section of Breast Surgery at Rigshospitalet, Copenhagen. Of these 324 participants enter the randomized controlled trial (RCT) and are randomized in a computer-generated sequence of 1:1 to the intervention (nurse-navigation) or control group (standard care). A total of 432 participants will enter an observational questionnaire study. All participants are followed for 1,5 years.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with breast cancer (i.e. prior to surgery), scheduled for breast cancer surgery at Section of Breast Surgery at Rigshospitalet, 18 years or above, Danish citizen, read, understand and speak Danish, female gender,signed written informed consent. Those who experience high psychological distress (score ≥ 7 on the distress thermometer) will enter the RCT whereas those who experience low psychological distress (score < 7 on the distress thermometer) will be followed in an observational questionnaire study.

Exclusion Criteria:

* no severe cognitive problems or dementia, no severe psychiatric disease requiring treatment, e.g. schizophrenia, alcohol or narcotic dependence,

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Distress | Change from baseline and to 6,12 months (mixed models)
  Distress Thermometer

SECONDARY OUTCOMES:
Distress | Change from baseline to 6 months
  Distress Thermometer
Distress | Change from baseline to 12 months
  Distress Thermometer
Distress | Change from baseline to 18 months
  Distress Thermometer
Depression | Change from baseline and to 3, 10, 18 weeks, 6,12,18 months (mixed models)
  The Patient Health Questionnaire (PHQ9)
Depression | Change from baseline and to 6 months
  The Patient Health Questionnaire (PHQ9)
Depression | Change from baseline and to 12 months
  The Patient Health Questionnaire (PHQ9)
Depression | Change from baseline and to 18 months
  The Patient Health Questionnaire (PHQ9)
Anxiety | Change from baseline and to 3, 10, 18 weeks, 6,12,18 months (mixed models)
  Generalized Anxiety Disorder (GAD7)
Anxiety | Change from baseline and to 6 months
  Generalized Anxiety Disorder (GAD7)
Anxiety | Change from baseline and to 12 months
  Generalized Anxiety Disorder (GAD7)
Anxiety | Change from baseline and to 18 months
  Generalized Anxiety Disorder (GAD7)
Health related quality of life summary index | Change from baseline and to 3, 10, 18 weeks, 6,12,18 months (mixed models)
  The Trial Outcome Index-Physical/Functional/Breast (TOI-PFB) score including Domains:
  * Physical well-being (PWB)
  * Functional wellbeing (FWB)
  * BC symptoms (BCS) from the Functional Assessment of Chronic Illness Therapy - Breast (FACT-B)
Health related quality of life summary index | Change from baseline and to 6 months
  The Trial Outcome Index-Physical/Functional/Breast (TOI-PFB) score including Domains:
  * Physical well-being (PWB)
  * Functional wellbeing (FWB)
  * BC symptoms (BCS) from the Functional Assessment of Chronic Illness Therapy - Breast (FACT-B)
Health related quality of life summary index | Change from baseline and to 12 months
  The Trial Outcome Index-Physical/Functional/Breast (TOI-PFB) score including Domains:
  * Physical well-being (PWB)
  * Functional wellbeing (FWB)
  * BC symptoms (BCS) from the Functional Assessment of Chronic Illness Therapy - Breast (FACT-B)
Health related quality of life summary index | Change from baseline and to 18 months
  The Trial Outcome Index-Physical/Functional/Breast (TOI-PFB) score including Domains:
  * Physical well-being (PWB)
  * Functional wellbeing (FWB)
  * BC symptoms (BCS) from the Functional Assessment of Chronic Illness Therapy - Breast (FACT-B)
Breast cancer related quality of life summary index | Change from baseline and to 3, 10, 18 weeks, 6,12,18 months (mixed models)
  BC symptoms (BCS) from the Functional Assessment of Chronic Illness Therapy - Breast (FACT-B)
Breast cancer related quality of life summary index | Change from baseline and to 6 months
  BC symptoms (BCS) from the Functional Assessment of Chronic Illness Therapy - Breast (FACT-B)
Breast cancer related quality of life summary index | Change from baseline and to 12 months
  BC symptoms (BCS) from the Functional Assessment of Chronic Illness Therapy - Breast (FACT-B)
Breast cancer related quality of life summary index | Change from baseline and to 18 months
  BC symptoms (BCS) from the Functional Assessment of Chronic Illness Therapy - Breast (FACT-B)
Functional related quality of life summary index | Change from baseline and to 3, 10, 18 weeks, 6,12,18 months (mixed models)
  Functional wellbeing (FWB) from the Functional Assessment of Chronic Illness Therapy - Breast (FACT-B)
Functional related quality of life summary index | Change from baseline and to 6 months
  Functional wellbeing (FWB) from the Functional Assessment of Chronic Illness Therapy - Breast (FACT-B)
Functional related quality of life summary index | Change from baseline and to 12 months
  Functional wellbeing (FWB) from the Functional Assessment of Chronic Illness Therapy - Breast (FACT-B)
Functional related quality of life summary index | Change from baseline and to 18 months
  Functional wellbeing (FWB) from the Functional Assessment of Chronic Illness Therapy - Breast (FACT-B)
Physical health related quality of life | Change from baseline and to 3, 10, 18 weeks, 6,12,18 months (mixed models)
  Physical well-being (PWB) from the Functional Assessment of Chronic Illness Therapy - Breast (FACT-B)
Physical health related quality of life | Change from baseline and to 6 months
  Physical well-being (PWB) from the Functional Assessment of Chronic Illness Therapy - Breast (FACT-B)
Physical health related quality of life | Change from baseline and to 12 months
  Physical well-being (PWB) from the Functional Assessment of Chronic Illness Therapy - Breast (FACT-B)
Physical health related quality of life | Change from baseline and to 18 months
  Physical well-being (PWB) from the Functional Assessment of Chronic Illness Therapy - Breast (FACT-B)
Social health related quality of life | Change from baseline and to 3, 10, 18 weeks, 6,12,18 months (mixed models)
  Social/Family well-being (SWB) from the Functional Assessment of Chronic Illness Therapy - Breast (FACT-B)
Social health related quality of life | Change from baseline and to 6 months
  Social/Family well-being (SWB) from the Functional Assessment of Chronic Illness Therapy - Breast (FACT-B)
Social health related quality of life | Change from baseline and to 12 months
  Social/Family well-being (SWB) from the Functional Assessment of Chronic Illness Therapy - Breast (FACT-B)
Social health related quality of life | Change from baseline and to 18 months
  Social/Family well-being (SWB) from the Functional Assessment of Chronic Illness Therapy - Breast (FACT-B)
Emotional health related quality of life | Change from baseline and to 3, 10, 18 weeks, 6,12,18 months (mixed models)
  Emotional well-being (EWB) from the Functional Assessment of Chronic Illness Therapy - Breast (FACT-B)
Emotional health related quality of life | Change from baseline and to 6 months
  Emotional well-being (EWB) from the Functional Assessment of Chronic Illness Therapy - Breast (FACT-B)
Emotional health related quality of life | Change from baseline and to 12 months
  Emotional well-being (EWB) from the Functional Assessment of Chronic Illness Therapy - Breast (FACT-B)
Emotional health related quality of life | Change from baseline and to 18 months
  Emotional well-being (EWB) from the Functional Assessment of Chronic Illness Therapy - Breast (FACT-B)
Self-efficacy | Change from baseline and to 6,12,18 months (mixed models)
  Patient Activation Measure (PAM)
Self-efficacy | Change from baseline and to 6 months
  Patient Activation Measure (PAM)
Self-efficacy | Change from baseline and to 12 months
  Patient Activation Measure (PAM)
Self-efficacy | Change from baseline and to 18 months
  Patient Activation Measure (PAM)
Fear of recurrence | 6 months
  Concerns About Recurrence Questionnaire (CARQ)
Fear of recurrence | 12 months
  Concerns About Recurrence Questionnaire (CARQ)
Fear of recurrence | 18 months
  Concerns About Recurrence Questionnaire (CARQ)
Pain in the breast surgery area (side of chest, armpit or arm) | Change from baseline and to 6,12,18 months (mixed models)
  Self-developed scale
Pain in the breast surgery area (side of chest, armpit or arm) | Change from baseline and to 6 months
  Self-developed scale
Pain in the breast surgery area (side of chest, armpit or arm) | Change from baseline and to 12 months
  Self-developed scale
Pain in the breast surgery area (side of chest, armpit or arm) | Change from baseline and to 18 months
  Self-developed scale
Neuropathy in the breast surgery area (side of chest, armpit or arm) | Change from baseline and to 6,12,18 months (mixed models)
  Self-developed scale
Neuropathy in the breast surgery area (side of chest, armpit or arm) | Change from baseline and to 6 months
  Self-developed scale
Neuropathy in the breast surgery area (side of chest, armpit or arm) | Change from baseline and to 12 months
  Self-developed scale
Neuropathy in the breast surgery area (side of chest, armpit or arm) | Change from baseline and to 18 months
  Self-developed scale
Sleep quality | Change from baseline and to 6,12,18 months (mixed models)
  Pittsburgh Sleep Quality Index (PSQI)
Sleep quality | Change from baseline and to 6 months
  Pittsburgh Sleep Quality Index (PSQI)
Sleep quality | Change from baseline and to 12 months
  Pittsburgh Sleep Quality Index (PSQI)
Sleep quality | Change from baseline and to 18 months
  Pittsburgh Sleep Quality Index (PSQI)
Cognitive function - Perceived cognitive impairments | Change from baseline and to 6,12,18 months (mixed models)
  Functional Assessment of Chronic Illness Therapy - Cognitive function (FACT-cog) - Sub-scale Perceived cognitive impairments
Cognitive function - Perceived cognitive impairments | Change from baseline and to 6 months
  Functional Assessment of Chronic Illness Therapy - Cognitive function (FACT-cog) - Sub-scale Perceived cognitive impairments
Cognitive function- Perceived cognitive impairments | Change from baseline and to 12 months
  Functional Assessment of Chronic Illness Therapy - Cognitive function (FACT-cog) - Sub-scale Perceived cognitive impairments
Cognitive function - Perceived cognitive impairments | Change from baseline and to 18 months
  Functional Assessment of Chronic Illness Therapy - Cognitive function (FACT-cog) - Sub-scale Perceived cognitive impairments
Cognitive function - Impact of Perceived cognitive impairments on quality of life | Change from baseline and to 6,12,18 months (mixed models)
  Functional Assessment of Chronic Illness Therapy - Cognitive function (FACT-cog) - Sub-scale - Impact of Perceived cognitive impairments on quality of life
Cognitive function - Impact of Perceived cognitive impairments on quality of life | Change from baseline and to 6 months
  Functional Assessment of Chronic Illness Therapy - Cognitive function (FACT-cog) - Sub-scale - Impact of Perceived cognitive impairments on quality of life
Cognitive function - Impact of Perceived cognitive impairments on quality of life | Change from baseline and to 12 months
  Functional Assessment of Chronic Illness Therapy - Cognitive function (FACT-cog) - Sub-scale - Impact of Perceived cognitive impairments on quality of life
Cognitive function - Impact of Perceived cognitive impairments on quality of life | Change from baseline and to 18 months
  Functional Assessment of Chronic Illness Therapy - Cognitive function (FACT-cog) - Sub-scale - Impact of Perceived cognitive impairments on quality of life
Cognitive function - Perceived cognitive abilities | Change from baseline and to 6,12,18 months (mixed models)
  Functional Assessment of Chronic Illness Therapy - Cognitive function (FACT-cog) - Sub-scale - Perceived cognitive abilities
Cognitive function - Perceived cognitive abilities | Change from baseline and to 6 months
  Functional Assessment of Chronic Illness Therapy - Cognitive function (FACT-cog) - Sub-scale - Perceived cognitive abilities
Cognitive function - Perceived cognitive abilities | Change from baseline and to 12 months
  Functional Assessment of Chronic Illness Therapy - Cognitive function (FACT-cog) - Sub-scale - Perceived cognitive abilities
Cognitive function - Perceived cognitive abilities | Change from baseline and to 18 months
  Functional Assessment of Chronic Illness Therapy - Cognitive function (FACT-cog) - Sub-scale - Perceived cognitive abilities
Need for support | Change from baseline and to 6,12,18 months (mixed models)
  Single self-developed items
Need for support | Change from baseline and to 6 months
  Single self-developed items
Need for support | Change from baseline and to 12 months
  Single self-developed items
Need for support | Change from baseline and to 18 months
  Single self-developed items
Health care costs | Cumulative from baseline to 18 months
  Costs will be obtained through registries on health care services and combined with information on health status using the 5Q-5D from the EuroQol Research Foundation's
Acceptability | 18 months
  Single self-developed items

OTHER OUTCOMES:
Social support | Baseline
  Modified Medical Outcomes Study Social Support Scale (MOS)

CONTACTS AND LOCATIONS:
Overall Officials: Pernille Bidstrup, PhD, Principal Investigator — Danish Cancer Society Research Center; Christoffer Johansen, DMSc, Principal Investigator — Rigshispitalet; Birgitte Mertz, RN, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bidstrup PE, Johansen C, Kroman N, Belmonte F, Duriaud H, Dalton SO, Andersen KG, Mertz B. Effect of a Nurse Navigation Intervention on Mental Symptoms in Patients With Psychological Vulnerability and Breast Cancer: The REBECCA Randomized Clinical Trial. JAMA Netw Open. 2023 Jun 1;6(6):e2319591. doi: 10.1001/jamanetworkopen.2023.19591. PMID 37351885